CLINICAL TRIAL: NCT01192919
Title: Clinical Registry Describing Treatment Reality and Therapy Modalities of Patients With Lung Cancer (NSCLC, SCLC and Neuroendocrine Tumors) Requiring Therapy.
Brief Title: Tumour Registry Lung Cancer (TLK)
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM TLK
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Lung Cancer
Keywords: bronchial carcinoma; registry; real life treatment; cohort study; NSCLC; SCLC; Germany
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Bronchogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with lung cancer: Patients with lung cancer requiring therapy

SUMMARY:
Overview of treatment reality in patients with bronchial carcinoma requiring systemic treatment and being treated by office-based oncologists in Germany.

DETAILED DESCRIPTION:
The TLK is a prospective, longitudinal, nation wide cohort study that collects data on the treatment reality of patients with NSCLC and SCLC. At inclusion, data in patient characteristics, comorbidities, tumor characteristics, biomarker testing and previous treatments are collected. During the course of observation data on all systemic treatments, radiotherapies, surgeries, and outcome are documented. Patients are followed until death or for a maximum of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed Small Cell Lung Cancer (SCLC), Non Small Lung Cancer (NSCLC) or neuroendocrine tumors receiving therapy
* written informed consent
* start of neoadjuvant, adjuvant or first-line therapy no longer than 4 weeks before informed consent

Exclusion Criteria:

* patients not receiving any systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with lung cancer requiring therapy
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2010-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Documentation of actually used therapy forms in bronchial carcinoma requiring treatment | 3 years per patient

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Werner Tessen, MD, Principal Investigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] von Verschuer U, Schnell R, Tessen HW, Eggert J, Binninger A, Spring L, Janicke M, Marschner N; TLK-Group (Tumour Registry Lung Cancer). Treatment, outcome and quality of life of 1239 patients with advanced non-small cell lung cancer - final results from the prospective German TLK cohort study. Lung Cancer. 2017 Oct;112:216-224. doi: 10.1016/j.lungcan.2017.07.031. Epub 2017 Sep 12. PMID 28916198
- [Result] Steffens CC, Elender C, Hutzschenreuter U, Dille S, Binninger A, Spring L, Janicke M, Marschner N; TLK-Group (Tumour Registry Lung Cancer). Treatment and outcome of 432 patients with extensive-stage small cell lung cancer in first, second and third line - Results from the prospective German TLK cohort study. Lung Cancer. 2019 Apr;130:216-225. doi: 10.1016/j.lungcan.2019.02.026. Epub 2019 Feb 25. Erratum In: Lung Cancer. 2019 Sep;135:236. doi: 10.1016/j.lungcan.2019.07.013. PMID 30885347